CLINICAL TRIAL: NCT01968642
Title: Educational Intervention to Reduce Outpatient Inappropriate Transthoracic Echocardiograms Ordered by Attending Physicians
Brief Title: Education and Feedback Intervention to Reduce Inappropriate Transthoracic Echocardiograms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rory Weiner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2011P001779 AME3
Record Dates: First submitted 2013-10-20; First posted 2013-10-24 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Inappropriate and Appropriate Transthoracic Echocardiograms
Keywords: Transthoracic echocardiograms; Appropriate Use Criteria; Medical Education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational Intervention (Experimental): Attending physicians in the intervention arm will receive the following multi-faceted educational intervention on transthoracic echocardiogram appropriateness: 1) a lecture at the beginning of the study period, which describes Appropriate USe Criteria (AUC) and highlights common clinical scenarios for which outpatient echocardiograms are ordered, 2) an electronic "pocket cared" via email that provides tips on appropriate ordering of echocardiograms, and 3) an individualized monthly feedback report that categorizes echocardiograms ordered over the preceding month. The feedback report will contain the number of echocardiograms ordered during the month and how many are classified as appropriate, inappropriate, or uncertain based on the 2011 AUC.
  Interventions: Behavioral: Educational Intervention
- Control Group (No Intervention): Attending physicians in the control arm will have their echocardiogram orders tracked and classified, but will not receive any feedback on their ordering behavior.

INTERVENTIONS:
Behavioral: Educational Intervention
  Arms: Educational Intervention

SUMMARY:
The utilization of transthoracic echocardiography in the United States has been increasing. This has resulted in increased costs to the healthcare system. In an effort to curb excessive utilization of this technology, the American College of Cardiology created Appropriate Use Criteria to help guide clinicians to use this diagnostic imaging modality more appropriately. The investigators previously showed that an educational intervention can reduce the rate of inappropriate echocardiograms ordered by physicians-in-training. It is unknown if such an intervention would be successful in attending, staff level of physicians. The investigators hypothesize that an educational and feedback intervention will reduce the rate of inappropriate outpatient transthoracic echocardiograms ordered by staff cardiologists and internal medicine physicians.

DETAILED DESCRIPTION:
In response to increasing utilization of echocardiography, the American Society of Echocardiography along with the American College of Cardiology released Appropriate Use Criteria (AUC) for transthoracic echocardiography (TTE) in 2007, and these have been subsequently updated in 2011. TTE ordering patterns have been evaluated and have shown that between 15-30% of TTE ordered are inappropriate. The highest rate of inappropriate TTE is found in the outpatient environment, where routine or "surveillance" studies are common. These studies have also found that internists and cardiologists order the majority of TTE. The investigators previously documented that an AUC-based educational and feedback intervention reduced the rate of inappropriate TTE by cardiology and internal medicine physicians-in-training. Whether this type of intervention can improve TTE ordering of attending level physicians is not known.

ELIGIBILITY:
Inclusion Criteria:

* Cardiology Attending physicians at Massachusetts General Hospital
* Primary care physicians at Massachusetts General Hospital

Exclusion Criteria:

* Physicians-in-training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Inappropriate transthoracic echocardiograms | 12 months
  Rate of inappropriate echocardiograms determined from a review of the electronic medical record.

SECONDARY OUTCOMES:
Rate of Appropriate transthoracic echocardiograms | 12 months
  Rate of appropriate transthoracic echocardiograms determined from a review of the electronic medical record.

OTHER OUTCOMES:
Clinical reasons for appropriate and inappropriate transthoracic echocardiograms | 12 months
  All echocardiograms will be classified according to the Appropriate Use Criteria (AUC). This will allow for determination of the most common clinical indications for both appropriate and inappropriate echocardiograms.

CONTACTS AND LOCATIONS:
Overall Officials: Rory B Weiner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bhatia RS, Milford CE, Picard MH, Weiner RB. An educational intervention reduces the rate of inappropriate echocardiograms on an inpatient medical service. JACC Cardiovasc Imaging. 2013 May;6(5):545-55. doi: 10.1016/j.jcmg.2013.01.010. Epub 2013 Apr 10. PMID 23582360
- [Derived] Dudzinski DM, Bhatia RS, Mi MY, Isselbacher EM, Picard MH, Weiner RB. Effect of Educational Intervention on the Rate of Rarely Appropriate Outpatient Echocardiograms Ordered by Attending Academic Cardiologists: A Randomized Clinical Trial. JAMA Cardiol. 2016 Oct 1;1(7):805-812. doi: 10.1001/jamacardio.2016.2232. PMID 27547895